CLINICAL TRIAL: NCT00640172
Title: Anemia in the Elderly
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stanley L Schrier, Professor of Medicine (Hematology), Emeritus, Stanford University
Other Study IDs: IRB-05112; SPO 36101 (Other: Stanford University); SU-01082008-967 (Other: Stanford University)
Record Dates: First submitted 2008-03-06; First posted 2008-03-21 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine and bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Anemic Elderly
- Non-anemic adults (non-elderly, without bone marrow biopsy)
- Non-anemic adults (non-elderly, with bone marrow biopsy)
- Non-anemic Elderly (control without bone marrow biopsy)
- Non-anemic Elderly (control, with bone marrow biopsy)

SUMMARY:
Eligible elderly men and women with anemia will undergo a full hematologic evaluation plus additional laboratory tests to determine the etiology of the anemia. In a subset of subjects, bone marrow aspirate and biopsies will be obtained for a planned analysis of erythroid progenitor and stem cells. Plasma; serum; and bone marrow samples will be will be compared to elderly non-anemic controls. Bone marrow samples will also be compared to non-anemic young controls (purchased).

DETAILED DESCRIPTION:
Eligible elderly men and women with anemia will undergo a full hematologic evaluation (blood sample for complete blood count, CBC) to determine the etiology of the anemia (eg, myelodysplastic syndrome). Peripheral smears; iron studies; serum creatinine; serum erythropoietin; reticulocyte count; vitamin B12; and folate levels may be obtained/conducted. When no etiology is identified (ie, "unexplained anemia"), additional laboratory tests will be performed which will include some or all of urinary hepcidin levels; plasma cytokine levels; serum soluble transferrin receptor; C-reactive protein; erythrocyte sedimentation rate; D-Dimer; neopterin level; tryptophan level; and blood for a cytokine profile that may include IL-1, IL-6, TNF-alpha, and VEGF levels. Serum; plasma; and nucleated peripheral blood cells may be banked for future DNA and other analyses. In a subset of those found to have either unexplained anemia (approximately 6 to 30 subjects) or anemia of chronic inflammation (approximately 6 to 30 subjects) , bone marrow aspirate and biopsies may be performed for a planned analysis of erythroid progenitor and stem cells in these populations. In addition, plasma and serum and bone marrow samples will be obtained from elderly non-anemic controls (approximately 6 to 30 subjects), and bone marrow samples will be purchased for non-anemic young controls (approximately 6 to 30 subjects) .

ELIGIBILITY:
INCLUSION CRITERIA: Anemic elderly :

* Age 65 or older
* Hemoglobin < 13 g/dL (men) or < 12 g/dL (women) on at least 2 occasions 30 days apart, with the most recent value within at least 14 days of enrollment into the study. In addition, if a CBC is drawn on the date of enrollment, hemoglobin must meet eligibility criteria in order for the patient to enroll.
* Outpatient at either the Stanford Health Care (SHC) Medical Center or VA Palo Alto Health Care System
* Independent/community living
* Ability to understand and the willingness to sign a written informed consent document
* Performance level ECOG 2 or better.

INCLUSION CRITERIA: Non-anemic elderly control, for blood and urine samples, with or without bone marrow biopsy

* Age 65 or older
* Hemoglobin ≥ 13 g/dL (men) or ≥ 12 g/dL (women) within at least 90 days of enrollment into the study
* Normal white blood cell and platelet counts
* Independent / community living
* Ability to understand and the willingness to sign a written informed consent document
* Performance level ECOG 2 or better
* Matched to UA population by gender and 10-year age strata (65 to < 75; 75 to < 85; 85 or older).

INCLUSION CRITERIA: Non-anemic adult control (non-elderly), for blood and urine samples, with bone marrow biopsy

* Age 20 to 35
* Hemoglobin ≥ 13 g/dL (men) or ≥ 12 g/dL (women) within at least 90 days of enrollment into the study
* Normal white blood cell and platelet counts
* Independent / community living
* Written informed consent obtained
* Performance level ECOG 2 or better

Inclusion Criteria: Non-anemic adult control (non-elderly), for blood and urine samples only

* Age 20 to 64
* Hemoglobin ≥ 13 g/dL (men) or ≥ 12 g/dL (women) within at least 90 days of enrollment into the study
* Normal white blood cell and platelet counts
* Independent / community living
* Written informed consent obtained
* Performance level ECOG 2 or better
* Will be recruited by the following age strata: 20 to < 35; 35 to < 50; 50 to < 65.

INCLUSION CRITERIA: Non-anemic adult control (non-elderly), with bone marrow biopsy

* Age 20 to 35
* Hemoglobin ≥ 13 g/dL (men) or ≥ 12 g/dL (women)

EXCLUSION CRITERIA: For all groups

* Substance abuse or mental health or other problems that would make compliance with the protocol unlikely
* Predicted mortality in less than 3 months, based on co-morbidities
* Known diagnosis of bone marrow disorder such as

  * Leukemia
  * Metastatic malignancy with bone marrow involvement
  * Myelodysplastic syndrome
  * Monoclonal gammopathy of undetermined significance (MGUS)
* On any erythropoiesis-stimulating agent in the prior 3 months
* Having received any red blood cell transfusion in the prior 3 months
* End stage renal disease as defined by the need for ongoing hemo or peritoneal dialysis
* Endstage liver disease as defined by the patient¡-s providers in the medical record
* A medical condition which would make participation risky
* On any other study requiring ongoing blood or marrow donation which would make additional blood or marrow collection risky to the subject

EXCLUSION CRITERIA: Additional, for healthy controls:

* History of active malignancy (except non-melanoma skin cancer), or radiation or chemotherapy for treatment of malignancy within the past 24 months
* HIV positivity
* Hepatitis B or Hepatitis C positivity
* Autoimmune disease (including lupus, RA, IBD)
* Known hematologic disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient elderly men and women (aged 65 years or older) with anemia, and corresponding elderly controls and adult non-elderly controls.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley L Schrier, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University School of Medicine, Stanford, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Price EA, Mehra R, Holmes TH, Schrier SL. Anemia in older persons: etiology and evaluation. Blood Cells Mol Dis. 2011 Feb 15;46(2):159-65. doi: 10.1016/j.bcmd.2010.11.004. Epub 2011 Jan 3. PMID 21208814